CLINICAL TRIAL: NCT02207270
Title: A Randomized Cost Minimization Analysis Comparing Same Day Discharge With Overnight Hospital Stay Following Elective and Low Risk Urgent Percutaneous Coronary Intervention.
Brief Title: Study Of Costs Realized After Percutaneous Coronary intervenTion Employing Same Day Discharge
Acronym: SOCRATES
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to meet projected enrollment
Sponsor: Trinity Health Michigan (Other)
Collaborators: Michigan Heart, PC (Other); Blue Cross Blue Shield of Michigan Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HSR-14-1479; 2033.11 (Other Grant/Funding Number: Blue Cross Blue Shield of Michigan Foundation)
Record Dates: First submitted 2014-07-28; First posted 2014-08-04 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Costs; Cost minimization; Percutaneous coronary intervention; Risk score; Same day discharge
MeSH Terms: conditions — Coronary Artery Disease | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomized clinical trail
Oversight: Data Monitoring Committee: No

ARMS (2):
- Same day discharge (Experimental): Patients who experienced uncomplicated PCI as well as an uncomplicated 6-hour observation period, will be randomly assigned to same day discharge.
  Interventions: Behavioral: Same day discharge
- Overnight stay standard care (Other): Patients who experienced uncomplicated PCI, as well as an uncomplicated 6-hour observation period, will be randomly assigned to an overnight stay, generally considered standard care.
  Interventions: Behavioral: Overnight Stay

INTERVENTIONS:
Behavioral: Same day discharge — Patients randomized to SDD will be discharged home on the day of their PCI, at least 6 hours following its completion. They will receive a follow up phone call from a study coordinator the next day and at 30 days to ascertain what costs (if any) were accrued and whether any adverse outcomes occurred.
  Other Names: SOCRATES
  Arms: Same day discharge
Behavioral: Overnight Stay — Patients who experienced uncomplicated PCI, as well as an uncomplicated 6-hour observation period, will be randomly assigned to an overnight stay, generally considered standard or routine care. Patients randomized to overnight stay will be discharged the following morning to receive a follow up phone call at 30 days to ascertain what costs (if any) were accrued and whether any adverse outcomes occurred.
  Other Names: Standard Care
  Arms: Overnight stay standard care

SUMMARY:
The purpose of this study is to determine whether the total costs of care associated with uncomplicated elective or low-risk urgent percutaneous coronary intervention (PCI) through 30-day follow up are lower among patients who are randomly assigned to same day discharge (SDD) or overnight hospital stay (ON).

DETAILED DESCRIPTION:
This is a prospective randomized clinical trial of same day discharge versus overnight stay for patients undergoing uncomplicated elective or low-risk urgent PCI with uncomplicated post-PCI recovery. The outcome is total cost accrued by patients from the time of index hospital presentation through 30-day post-PCI follow-up.

Conduct of PCI procedures and provision of post-PCI care will be in accordance with routine institutional practices and will not be protocol-driven.

Consented patients will be assigned to SDD or ON stay using a block randomization schedule. Randomization will occur once the patient has completed an uncomplicated 6-hour post PCI observation period.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients who undergo elective or low-risk, (i.e., in the setting of unstable angina but not non-ST segment elevation myocardial infarction) urgent PCI.
* No sociodemographic factors that would preclude SDD (prohibitive factors include no family member/friend available to remain with patient until nurse phone call the following day, no working phone, no reliable transportation, home > 60 minutes from medical infrastructure, unable to obtain/pay for medications).
* PCI procedures performed between 08/04/14 and 08/03/16.
* Short term risk of in-hospital death, transfusion or contrast-induced nephropathy during the index hospitalization at or below 1% using Blue Cross Blue Shield of Michigan Cardiovascular Consortium (BMC2) PCI registry risk prediction models.
* No in-lab complications (prolonged angina, acute closure, no reflow, significant or untreated dissection, vessel perforation, side branch occlusion, rescue glycoprotein IIb/IIIa inhibitor use, ventricular tachycardia or fibrillation requiring cardioversion/defibrillation, tamponade, pulmonary edema, stroke or transient ischemic attack, shock).
* Contrast Volume/Calculated Creatinine Clearance ratio < 3
* No recurrent chest pain, shortness of breath, hemodynamic instability, bleeding or vascular complications during 6 hours in recovery area post-PCI

Exclusion Criteria:

* Use of rotational atherectomy
* Use of a glycoprotein IIb/IIIa inhibitor infusion post-PCI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-08-11 (Actual); Primary Completion 2015-09-01 (Actual); Study Completion 2015-09-01 (Actual)

PRIMARY OUTCOMES:
Total costs from a modified societal perspective | Index hospital admission to 30-days post-PCI
  Costs will be determined from a modified societal perspective (physician labor, office visit and outpatient drug costs will not be included) and will be reported in 2014 dollars.

SECONDARY OUTCOMES:
Total costs from a 3rd party payer perspective | Index hospital admission to 30-days post-PCI
  Costs will be determined from a from a 3rd party payer perspective (physician labor, office visit and outpatient drug costs will also be included) and will be reported in 2014 dollars.
Adverse clinical outcomes | Index hospital admission to 30-days post-PCI
  Includes death, myocardial infarction, stroke, unplanned cardiac catheterization or coronary revascularization, vascular or hemorrhagic complications.
Rehospitalization | From discharge through 30-day post-PCI
  Inclusive of rehospitalization for any reason.

CONTACTS AND LOCATIONS:
Overall Officials: Herbert D. Aronow, MD, MPH, Principal Investigator — Michigan Heart, PC
Locations (2):
- United States (2):
  - Saint Joseph Mercy Health System, St. Joseph Mercy [Hospital] Ann Arbor, Cardiac Catheterization Laboratory, Ypsilanti, Michigan
  - Saint Jospeh Mercy Health System, St. Joseph Mercy [Hospital] Ann Arbor, Cardiac Catheterization Laboratory, Ypsilanti, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdelaal E, Rao SV, Gilchrist IC, Bernat I, Shroff A, Caputo R, Costerousse O, Pancholy SB, Bertrand OF. Same-day discharge compared with overnight hospitalization after uncomplicated percutaneous coronary intervention: a systematic review and meta-analysis. JACC Cardiovasc Interv. 2013 Feb;6(2):99-112. doi: 10.1016/j.jcin.2012.10.008. Epub 2013 Jan 23. PMID 23352820
- [Background] Amin AP, Marso SP, Rao SV, Messenger J, Chan PS, House J, Kennedy K, Robertus K, Cohen DJ, Mahoney EM. Cost-effectiveness of targeting patients undergoing percutaneous coronary intervention for therapy with bivalirudin versus heparin monotherapy according to predicted risk of bleeding. Circ Cardiovasc Qual Outcomes. 2010 Jul;3(4):358-65. doi: 10.1161/CIRCOUTCOMES.110.957290. Epub 2010 May 20. PMID 20488917
- [Background] Antman EM, Cohen M, Bernink PJ, McCabe CH, Horacek T, Papuchis G, Mautner B, Corbalan R, Radley D, Braunwald E. The TIMI risk score for unstable angina/non-ST elevation MI: A method for prognostication and therapeutic decision making. JAMA. 2000 Aug 16;284(7):835-42. doi: 10.1001/jama.284.7.835. PMID 10938172
- [Background] Barber JA, Thompson SG. Analysis of cost data in randomized trials: an application of the non-parametric bootstrap. Stat Med. 2000 Dec 15;19(23):3219-36. doi: 10.1002/1097-0258(20001215)19:233.0.co;2-p. PMID 11113956
- [Background] Brayton KM, Patel VG, Stave C, de Lemos JA, Kumbhani DJ. Same-day discharge after percutaneous coronary intervention: a meta-analysis. J Am Coll Cardiol. 2013 Jul 23;62(4):275-85. doi: 10.1016/j.jacc.2013.03.051. Epub 2013 Apr 23. PMID 23623905
- [Background] Chambers CE, Dehmer GJ, Cox DA, Harrington RA, Babb JD, Popma JJ, Turco MA, Weiner BH, Tommaso CL; Society for Cardiovascular Angiography and Interventions. Defining the length of stay following percutaneous coronary intervention: an expert consensus document from the Society for Cardiovascular Angiography and Interventions. Endorsed by the American College of Cardiology Foundation. Catheter Cardiovasc Interv. 2009 Jun 1;73(7):847-58. doi: 10.1002/ccd.22100. PMID 19425053
- [Background] Dangas GD, Claessen BE, Mehran R, Xu K, Fahy M, Parise H, Henriques JP, Ohman EM, White HD, Stone GW. Development and validation of a stent thrombosis risk score in patients with acute coronary syndromes. JACC Cardiovasc Interv. 2012 Nov;5(11):1097-105. doi: 10.1016/j.jcin.2012.07.012. PMID 23174632
- [Background] Farooq V, van Klaveren D, Steyerberg EW, Meliga E, Vergouwe Y, Chieffo A, Kappetein AP, Colombo A, Holmes DR Jr, Mack M, Feldman T, Morice MC, Stahle E, Onuma Y, Morel MA, Garcia-Garcia HM, van Es GA, Dawkins KD, Mohr FW, Serruys PW. Anatomical and clinical characteristics to guide decision making between coronary artery bypass surgery and percutaneous coronary intervention for individual patients: development and validation of SYNTAX score II. Lancet. 2013 Feb 23;381(9867):639-50. doi: 10.1016/S0140-6736(13)60108-7. PMID 23439103
- [Background] Gilchrist IC, Rhodes DA, Zimmerman HE. A single center experience with same-day transradial-PCI patients: a contrast with published guidelines. Catheter Cardiovasc Interv. 2012 Mar 1;79(4):583-7. doi: 10.1002/ccd.23159. Epub 2011 May 13. PMID 21542123
- [Background] Glaser R, Gertz Z, Matthai WH, Wilensky RL, Weiner M, Kolansky D, Hirshfeld J Jr, Herrmann H. Patient satisfaction is comparable to early discharge versus overnight observation after elective percutaneous coronary intervention. J Invasive Cardiol. 2009 Sep;21(9):464-7. PMID 19726820
- [Background] Gurm HS, Dixon SR, Smith DE, Share D, Lalonde T, Greenbaum A, Moscucci M; BMC2 (Blue Cross Blue Shield of Michigan Cardiovascular Consortium) Registry. Renal function-based contrast dosing to define safe limits of radiographic contrast media in patients undergoing percutaneous coronary interventions. J Am Coll Cardiol. 2011 Aug 23;58(9):907-14. doi: 10.1016/j.jacc.2011.05.023. PMID 21851878
- [Background] Gurm HS, Seth M, Kooiman J, Share D. A novel tool for reliable and accurate prediction of renal complications in patients undergoing percutaneous coronary intervention. J Am Coll Cardiol. 2013 Jun 4;61(22):2242-8. doi: 10.1016/j.jacc.2013.03.026. PMID 23721921
- [Background] Heyde GS, Koch KT, de Winter RJ, Dijkgraaf MG, Klees MI, Dijksman LM, Piek JJ, Tijssen JG. Randomized trial comparing same-day discharge with overnight hospital stay after percutaneous coronary intervention: results of the Elective PCI in Outpatient Study (EPOS). Circulation. 2007 May 1;115(17):2299-306. doi: 10.1161/CIRCULATIONAHA.105.591495. Epub 2007 Apr 9. PMID 17420341
- [Background] Jabara R, Gadesam R, Pendyala L, Chronos N, Crisco LV, King SB, Chen JP. Ambulatory discharge after transradial coronary intervention: Preliminary US single-center experience (Same-day TransRadial Intervention and Discharge Evaluation, the STRIDE Study). Am Heart J. 2008 Dec;156(6):1141-6. doi: 10.1016/j.ahj.2008.07.018. Epub 2008 Oct 9. PMID 19033010
- [Background] Khatri S, Webb JG, Carere RG, Amis A, Woolcott J, Chugh S, Humphries KH. Safety and cost benefit of same-day discharge after percutaneous coronary intervention. Am J Cardiol. 2002 Aug 15;90(4):425-7. doi: 10.1016/s0002-9149(02)02504-3. No abstract available. PMID 12161237
- [Background] Kim M, Muntner P, Sharma S, Choi JW, Stoler RC, Woodward M, Mann DM, Farkouh ME. Assessing patient-reported outcomes and preferences for same-day discharge after percutaneous coronary intervention: results from a pilot randomized, controlled trial. Circ Cardiovasc Qual Outcomes. 2013 Mar 1;6(2):186-92. doi: 10.1161/CIRCOUTCOMES.111.000069. Epub 2013 Mar 12. PMID 23481528
- [Background] Koch KT, Piek JJ, Prins MH, de Winter RJ, Mulder K, Lie KI, Tijssen JG. Triage of patients for short term observation after elective coronary angioplasty. Heart. 2000 May;83(5):557-63. doi: 10.1136/heart.83.5.557. PMID 10768908
- [Background] Mehran R, Aymong ED, Nikolsky E, Lasic Z, Iakovou I, Fahy M, Mintz GS, Lansky AJ, Moses JW, Stone GW, Leon MB, Dangas G. A simple risk score for prediction of contrast-induced nephropathy after percutaneous coronary intervention: development and initial validation. J Am Coll Cardiol. 2004 Oct 6;44(7):1393-9. doi: 10.1016/j.jacc.2004.06.068. PMID 15464318
- [Background] Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. No abstract available. PMID 21670242
- [Background] Mehta SK, Frutkin AD, Lindsey JB, House JA, Spertus JA, Rao SV, Ou FS, Roe MT, Peterson ED, Marso SP; National Cardiovascular Data Registry. Bleeding in patients undergoing percutaneous coronary intervention: the development of a clinical risk algorithm from the National Cardiovascular Data Registry. Circ Cardiovasc Interv. 2009 Jun;2(3):222-9. doi: 10.1161/CIRCINTERVENTIONS.108.846741. Epub 2009 May 8. PMID 20031719
- [Background] Moussa I, Hermann A, Messenger JC, Dehmer GJ, Weaver WD, Rumsfeld JS, Masoudi FA. The NCDR CathPCI Registry: a US national perspective on care and outcomes for percutaneous coronary intervention. Heart. 2013 Mar;99(5):297-303. doi: 10.1136/heartjnl-2012-303379. Epub 2013 Jan 15. PMID 23322530
- [Background] Moscucci M, Rogers EK, Montoye C, Smith DE, Share D, O'Donnell M, Maxwell-Eward A, Meengs WL, De Franco AC, Patel K, McNamara R, McGinnity JG, Jani SM, Khanal S, Eagle KA. Association of a continuous quality improvement initiative with practice and outcome variations of contemporary percutaneous coronary interventions. Circulation. 2006 Feb 14;113(6):814-22. doi: 10.1161/CIRCULATIONAHA.105.541995. Epub 2006 Feb 6. PMID 16461821
- [Background] Patel M, Kim M, Karajgikar R, Kodali V, Kaplish D, Lee P, Moreno P, Krishnan P, Sharma SK, Kini AS. Outcomes of patients discharged the same day following percutaneous coronary intervention. JACC Cardiovasc Interv. 2010 Aug;3(8):851-8. doi: 10.1016/j.jcin.2010.05.010. PMID 20723858
- [Background] Peterson ED, Dai D, DeLong ER, Brennan JM, Singh M, Rao SV, Shaw RE, Roe MT, Ho KK, Klein LW, Krone RJ, Weintraub WS, Brindis RG, Rumsfeld JS, Spertus JA; NCDR Registry Participants. Contemporary mortality risk prediction for percutaneous coronary intervention: results from 588,398 procedures in the National Cardiovascular Data Registry. J Am Coll Cardiol. 2010 May 4;55(18):1923-32. doi: 10.1016/j.jacc.2010.02.005. PMID 20430263
- [Background] Pinto DS, Stone GW, Shi C, Dunn ES, Reynolds MR, York M, Walczak J, Berezin RH, Mehran R, McLaurin BT, Cox DA, Ohman EM, Lincoff AM, Cohen DJ; ACUITY (Acute Catheterization and Urgent Intervention Triage Strategy) Investigators. Economic evaluation of bivalirudin with or without glycoprotein IIb/IIIa inhibition versus heparin with routine glycoprotein IIb/IIIa inhibition for early invasive management of acute coronary syndromes. J Am Coll Cardiol. 2008 Nov 25;52(22):1758-68. doi: 10.1016/j.jacc.2008.08.021. PMID 19022155
- [Background] Popescu AM, Weintraub WS. Outpatient percutaneous coronary interventions: hospital and health system costs saving while maintaining patient safety. JACC Cardiovasc Interv. 2010 Oct;3(10):1020-1. doi: 10.1016/j.jcin.2010.09.001. No abstract available. PMID 20965459
- [Background] Rao SC, Chhatriwalla AK, Kennedy KF, Decker CJ, Gialde E, Spertus JA, Marso SP. Pre-procedural estimate of individualized bleeding risk impacts physicians' utilization of bivalirudin during percutaneous coronary intervention. J Am Coll Cardiol. 2013 May 7;61(18):1847-52. doi: 10.1016/j.jacc.2013.02.017. Epub 2013 Mar 7. PMID 23500304
- [Background] Rao SV, Kaltenbach LA, Weintraub WS, Roe MT, Brindis RG, Rumsfeld JS, Peterson ED. Prevalence and outcomes of same-day discharge after elective percutaneous coronary intervention among older patients. JAMA. 2011 Oct 5;306(13):1461-7. doi: 10.1001/jama.2011.1409. PMID 21972308
- [Background] Rinfret S, Kennedy WA, Lachaine J, Lemay A, Rodes-Cabau J, Cohen DJ, Costerousse O, Bertrand OF. Economic impact of same-day home discharge after uncomplicated transradial percutaneous coronary intervention and bolus-only abciximab regimen. JACC Cardiovasc Interv. 2010 Oct;3(10):1011-9. doi: 10.1016/j.jcin.2010.07.011. PMID 20965458
- [Background] Rothwell PM, Giles MF, Flossmann E, Lovelock CE, Redgrave JN, Warlow CP, Mehta Z. A simple score (ABCD) to identify individuals at high early risk of stroke after transient ischaemic attack. Lancet. 2005 Jul 2-8;366(9479):29-36. doi: 10.1016/S0140-6736(05)66702-5. PMID 15993230
- [Background] Waksman R, Barbash IM. The appropriate use of risk scores. JACC Cardiovasc Interv. 2012 Nov;5(11):1106-7. doi: 10.1016/j.jcin.2012.08.007. No abstract available. PMID 23174633
- [Background] Yeh RW, Normand SL, Wolf RE, Jones PG, Ho KK, Cohen DJ, Cutlip DE, Mauri L, Kugelmass AD, Amin AP, Spertus JA. Predicting the restenosis benefit of drug-eluting versus bare metal stents in percutaneous coronary intervention. Circulation. 2011 Oct 4;124(14):1557-64. doi: 10.1161/CIRCULATIONAHA.111.045229. Epub 2011 Sep 6. PMID 21900079
- [Background] Ziakas AA, Klinke BP, Mildenberger CR, Fretz DE, Williams EM, Kinloch FR, Hilton j GJ. Safety of same-day-discharge radial percutaneous coronary intervention: a retrospective study. Am Heart J. 2003 Oct;146(4):699-704. doi: 10.1016/S0002-8703(03)00258-8. PMID 14564326
- [Background] Ziakas A, Klinke P, Fretz E, Mildenberger R, Williams MB, Siega AD, Kinloch RD, Hilton JD. Same-day discharge is preferred by the majority of the patients undergoing radial PCI. J Invasive Cardiol. 2004 Oct;16(10):562-5. PMID 15505350